CLINICAL TRIAL: NCT03351179
Title: Predictors and Outcomes of Hospitalized Heart Failure With Preserved Ejection Fraction Among Patients With First Acute Myocardial Infarction After Reperfusion Treatments
Brief Title: Predictors and Outcomes of In-hospital HFpEF in AMI Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xiangjun Yang (Other)
Responsible Party: Sponsor-Investigator, Xiangjun Yang, Director, department of cardiology, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Other Study IDs: FirstSoochowU
Record Dates: First submitted 2017-11-04; First posted 2017-11-22 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Acute Myocardial Infarction; Heart Failure With Preserved Ejection Fraction; Predictor; Prognosis
Keywords: Heart Failure with Preserved Ejection Fraction; Acute MyocAcute Myocardial Infarction; Predictive factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AMI patients with HFpEF
  Interventions: Combination Product: clinical characteristics, previous history, laboratory bio-markers, echocardiographic measurements, angiographic findings,clinical outcomes
- AMI patients without HF
  Interventions: Combination Product: clinical characteristics, previous history, laboratory bio-markers, echocardiographic measurements, angiographic findings,clinical outcomes

INTERVENTIONS:
Combination Product: clinical characteristics, previous history, laboratory bio-markers, echocardiographic measurements, angiographic findings,clinical outcomes — The differences of data(clinical characteristics, history, laboratory biomarkers, echocardiographic measurements, angiographic characteristics and clinical outcomes) in two groups were conducted. The differences between two groups were compared (clinical characteristics, history, laboratory biomarkers, echocardiographic measurements, angiographic characteristics and clinical outcomes) in two groups were compared, and then found the risk factors. Following,the incidence of clinical outcomes and mortality were compared. Then, univariate logistic regression and multivariate logistic regression analysis adjusted for significant risk factors were performed to find out the independent predictive factors. Finally, the ROC was constructed, and the area was evaluated to assess the predicted probability of regression model.

SUMMARY:
This retrospective observation is to investigate the incidence,clinical outcomes and prognosis of hospitalized heart failure with preserved ejection fraction (HFpEF) in patients with acute myocardial infarction(AMI).

DETAILED DESCRIPTION:
1. Patients with first AMI undergoing primary percutaneous coronary intervention (PCI) in our hospital since January 2013 were retrospectively evaluated. The enrolled subjects were divided into two groups (AMI patients with HFpEF and AMI patients without HF).
2. The investigator collected the clinical data of participants' demographics (age, sex), previous history,risk factors for AMI (hypertension, hyperlipidemia, diabetes mellitus, smoking and stroke), laboratory biomarkers, echocardiographic measurements, clinical characteristics,medical procedures and treatments, as well as in-hospital complications.
3. Two sub-investigators independently analyzed these data by using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* First AMI patients undergoing PCI with HFpEF or without HF.

Exclusion Criteria:

* First AMI patients with heart failure with reduced ejection fraction.
* First AMI patients with severe inflammatory diseases, valvular heart disease, non-cardiac caused symptoms, serious hepatic and renal failure, congenital cardiomyopathy,or pericardial diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AMI patients with HFpEF: First AMI subjects undergoing PCI with a diagnosis of HFpEF.
  AMI patients without HF: First AMI subjects undergoing PCI without a diagnosis of HF.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Risk factors of incident in-hospital HFpEF | Outcome measure will be assessed at discharge, and data will be reported through study completion, an average of 1 year.

SECONDARY OUTCOMES:
Clinical prognosis in patients with HFpEF | Outcome measure will be assessed at discharge, and data will be reported through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangjun Yang, PhD, Principal Investigator — First Affiliated Hospital of Soochow University
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided